CLINICAL TRIAL: NCT05517824
Title: Efficacy and Safety of the Micro-insulated Needle Radiofrequency Device for Reduction of Submental Fat
Brief Title: Needle Radiofrequency Treatment for Submental Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jung-Won Shin, Associate Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: B-2012-655-001
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: prospective, single-blinded, pre-post comparative study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-treatment (Active Comparator): After a single treatment using a microinsulated needle RF device
  Interventions: Procedure: microinsulated needle radiofrequency
- Pre-treatment (Baseline) (No Intervention)

INTERVENTIONS:
Procedure: microinsulated needle radiofrequency — A single treatment using a microinsulated needle radiofrequency device
  Arms: Post-treatment

SUMMARY:
The investigators aimed to evaluate the efficacy and safety of a fractional radiofrequency device with a micro-insulated needle to reduce submental fat.

ELIGIBILITY:
Inclusion Criteria:

* Patients with excess submental fat on a grade of 1~4, as assessed by the Physician-Assisted Submental Fat Rating Scale

Exclusion Criteria:

* mental impairment, infectious disease
* history of keloid development
* pregnancy, pacemaker
* use of anticoagulants
* undergoing a facelift procedure within the prior 6 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Physician-Assisted Submental Fat Rating Scale score from 0 (nothing) to 4 (very severe) | 1 month after the treatment
  submental fat rating by an independent investigator

SECONDARY OUTCOMES:
submental fat volume (cc) | 1 month after the treatment
  fat volume quantified with a three-dimensional camera
patient satisfaction score from 0 (not satisfied) to 10 (most satisfied) | 1 month after the treatment
  patient's satisfaction score for reduction of submental fat
any adverse effects at any time during or after treatment | assessed through study completion, an average of 2 months
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hun Huh, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim BR, Kim M, Kim JW, Shin JW, Na JI, Huh CH. Efficacy and Safety of the Micro-insulated Needle Radiofrequency Device for Reduction of Submental Fat. Dermatol Surg. 2023 Apr 1;49(4):389-394. doi: 10.1097/DSS.0000000000003723. Epub 2023 Feb 10. PMID 36799883